CLINICAL TRIAL: NCT00499824
Title: GIANT: General Practitioner Implementation in Asia of Normoglycaemic Targets
Acronym: GIANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Diabetes Institute, Australia (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Assoc Prof Jonathan Shaw & Professor Paul Zimmet, Baker IDI Heart and Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IDI Project 4/2006
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Management guidelines; Efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Medical Practitioners who receive education on diabetes management following the guidelines of the International Diabetes Federation Western Pacific Region
  Interventions: Behavioral: Education of general practitioners on the IDF-WPR guidelines
- 2 (No Intervention): Medical practitioners who follow standard practice for management of their patients with type 2 diabetes

INTERVENTIONS:
Behavioral: Education of general practitioners on the IDF-WPR guidelines — The intervention will comprise an educational program on the guidelines for GPs, and will be carried out by the national coordinating centre in each country, based on a template provided by the international coordinating centre (International Diabetes Institute, Australia). This will involve:
  an initial educational symposium and a follow-up continuing medical education symposium at 3 months; paper or electronic reminders of the guidelines sent to GPs every 3 months; desktop reminder cards with guideline algorithms; insertion of a flowsheet (diabetes action plan) into the patient's medical notes by the study nurse; provision of each patient with a "diabetes passport" to be held by the patient.
  Arms: 1

SUMMARY:
To test whether the International Diabetes Federation - Western Pacific Region (IDF-WPR) Guidelines are more effective than standard practices in primary care (general practitioner) clinics for the management of type 2 diabetes mellitus (T2DM) in Asia. A 12-month multinational multicentre prospective cluster randomisation clinical trial within a primary care setting, with 2 parallel treatment arms: diabetes management using IDF-WPR guidelines versus standard clinic practices. 400 subjects will be recruited from 100 sites (4 subjects per site) in ten Asian countries (China, Hong Kong, Indonesia, Korea, Malaysia, Philippines, Singapore, Taiwan, Thailand and Vietnam).

DETAILED DESCRIPTION:
Description of intervention(s) / exposure and control treatment: This is a prospective multinational, multicentre, cluster-randomised study conducted within the primary care setting, with two parallel treatment arms: standard clinical practice versus education on diabetes management using International Diabetes Federation - Western Pacific Region (IDF-WPR) "Type 2 diabetes practical targets and treatments". The study duration will be 12 months.

100 General Practitioners (GPs) (10 per country) will be randomised to receive education on the IDF-WPR guidelines or to receive no trial-related education.

* GPs in both groups will be required to recruit 4 of their own patients meeting the eligibility criteria. The complete entry criteria are detailed in a following section.
* GPs in both groups will manage the recruited patients according to their own clinical judgement. Frequency of patient visits to the GP's clinic will be determined by the GP. All medication prescribed by the GPs should already be registered in the participating countries.
* Blood sampling of patients will be required at Study Visit 1 (Screening/Baseline), Study Visit 2 (month 6) and Study Visit 3 (month 12).

The intervention will comprise an educational program on the guidelines for GPs, and will be carried out by the national coordinating centre in each country, based on a template provided by the international coordinating centre (International Diabetes Institute, Australia). The educational program for the GPs randomised to the intervention arm will:

1. Combine didactic and interactive sessions.
2. Involve opinion leaders, i.e. the national lead investigator
3. Aim to resolve barriers to practical implementation of guidelines already identified from previous studies (e.g. discuss starting insulin)
4. Present the evidence for the guidelines.
5. Highlight any conflicts between the guidelines and local prescribing regulations, and confirm the need to follow the local prescribing regulations in these instances
6. Involve an initial educational symposium and a follow-up continuing medical education symposium at 3 months

Organisational changes to improve guideline adherence for the study will include:

1. Paper or electronic reminders of the guidelines will be sent to GPs every 3 months.
2. Desktop reminders cards with key guideline algorithms.
3. Insertion of a flowsheet (diabetes action plan) into the patient's medical notes by the study nurse (at the time of review of the practitioner's baseline HbA1c utilisation).

Patient-centred approaches to improve guideline adherence for the study will include:

1. Encouragement and empowerment of patients to ask questions of the treating practitioners
2. Provision of each patient with a "diabetes passport" to be held by the patient, to encourage discussion between the patient and practitioner and also recording of results of medical examinations. This will be provided at the baseline visit to the national coordinating centre.

ELIGIBILITY:
INCLUSION CRITERIA

* Men or women who are 30 to 75 years of age (inclusive) at Study Visit 1.
* Clinical diagnosis of type 2 diabetes (defined according to IDF Guidelines) for a minimum of 6 months prior to Study Visit 1
* Patients for whom the GP is the primary medical provider of diabetes care and for whom referral to another doctor for diabetes care is not anticipated within 3 months of Study Visit 1
* Patients who give informed consent to participate.

EXCLUSION CRITERIA

* Patients with type 1 diabetes mellitus
* Patients with any previous episode of ketoacidosis
* Patients who required chronic use (>/= 6 months) of insulin at any time in the past, with the exception of females during pregnancy
* Patients receiving insulin treatment at Study Visit 1 or within the previous 6 months, with the exception of patients who received short-term treatment (= 7 days) with insulin to maintain glycaemic control for an acute event (e.g. hospitalisation or medical procedure/intervention, infection or trauma).
* Treatment with glucocorticoid at Study Visit 1 or within the previous 6 months, with the exception of topical or inhaled glucocorticoid
* Females who are pregnant or considering pregnancy or stopping contraception within the course of the study
* Patients with end-stage renal disease, defined as glomerular filtration rate (GFR) by the MDRD (Modification of Diet in Renal Disease) formula < 15 ml/min/1.73 m2, or on renal replacement therapy with haemodialysis, peritoneal dialysis or renal transplant.
* Patients with psychiatric disease, active drug or alcohol abuse or other cognitive impairment that may interfere with treatment compliance.
* Receipt of any investigational drug within 30 days of Study Visit 1.
* Patients receiving diabetes care from another doctor (specialist endocrinologist, general physician, or another GP) Other eligibility criteria considerations The HbA1c at entry for newly recruited patients will be monitored centrally. If there is a significant risk that more than 25% of the total study population will have a baseline HbA1c </= 6.5%, then recruitment of subsequent patients will be restricted to those with HbA1c > 6.5%.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline in subjects with baseline HbA1c >/=6.5% | 6 months

SECONDARY OUTCOMES:
HbA1c, FPG, BP, lipids; hypoglycemic events; health care use; number of GP HbA1c measurements; number of treatment escalations; adverse events; barriers to guideline implementation; determine if study patients are representative of GP's diabetic practice | 6 & 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan E Shaw, MD MRCP FRACP, Principal Investigator — International Diabetes Institute, Australia
Locations (10):
- China (2):
  - Department of Medicine & Therapeutics, Prince of Wales Hospital, The Chinese University of Hong Kong, Shatin, Hong Kong
  - Department of Endocrinology & Metabolism, Peking University People's Hospital, Beijing
- Diabetes and Nutrition Center, Dr. Soetomo Teaching Hospital - Airlangga University,, Surabaya, Indonesia
- School of Medicine and Health Sciences, Monash University House, Johor Bahru, Malaysia
- Section of Endocrinology, Diabetes and Metabolism, Department of Medicine, University of the Philippines College of Medicine, Manila, Philippines
- Diabetes, Lipid and Endocrine Practice, Gleneagles Medical Centre, Singapore, Singapore
- Department of Endocrinology & Metabolism, Kangnam St. Mary's Hospital, The Catholic University of Medicine, Seoul, South Korea
- Dept of Medical Research and Education, Taipei Veterans General Hospital,, Taipei, Taiwan
- Diabetes and Endocrinology Unit, Department of Medicine, Rajavithi Hospital,, Bangkok, Thailand
- National Hospital of Endocrinology,, Hanoi, Dongda District, Vietnam